CLINICAL TRIAL: NCT03579485
Title: An Observational Retrospective Database Analysis to Evaluate Raltegravir Based-regimens, Including NUC-sparing Regimens, in Aged HIV Patients.(RalAge)
Acronym: RalAge2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Policlinico Umberto I (Other)
Responsible Party: Principal Investigator, Gabriella D'Ettorre, Professor, Azienda Policlinico Umberto I
Other Study IDs: APUmbertoI RalAge2
Record Dates: First submitted 2018-06-26; First posted 2018-07-06 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Hiv
Keywords: raltegravir; naive; Aging
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- aging HIV positive patients: HIV-1 infected patients, aged ≥ 60 years old, naive patients receiving raltegravir based-regimen, including Nuc-sparing regimens or experienced patients with virological suppression (HIV-1 RNA<50 copies) who had switched from any antiretroviral drug to raltegravir-based regimens (including Nuc-sparing regimens) because of toxicity, convenience or other reasons.

SUMMARY:
This is an observational retrospective cohort in real world to describe RAL data, including NUC-sparing regimens, in aged HIV patients. It is a phase IV study.

90 patients will be enrolled from the Department of Public Health and Infectious Diseases of "Sapienza" University of Rome.

In this retrospective analysis all naïve patients on raltegravir-based regimens and all patients switched to raltegravir-based regimens will be considered.

DETAILED DESCRIPTION:
Antiretroviral therapy has changed the natural history of HIV infection. However, antiretroviral therapy must be maintained for life. Its potential long-term adverse effects may interact synergistically with the ageing process, resulting in a higher incidence of comorbidities. The increasing number of non-antiretroviral drugs used to treat comorbidities may also place the patient at a higher risk of clinically meaningful interactions. Nowadays, efficacy is well demonstrated by all antiretroviral drugs compared with previous times. In fact a substantial number of HIV-infected patients from areas where antiretroviral therapy is widely available have achieved sustained suppression of plasma HIV replication. In contrast, the contributions of antiretroviral therapy to the development and progression of comorbidities and to the risk of potentially severe interactions have gained increasing importance as HIV-infected patients are getting older. More than half of HIV-infected patients aged ≥ 50 years have been reported to suffer from two or more concomitant comorbidities. In some of these patients, maintenance of antiretroviral therapy with combinations including NRTIs or PIs may be challenging (1). Data on ageing HIV patients under antiretroviral therapy are lacking.

RAL is considered one of the better-tolerated antiretroviral medications, due to limited side effects and few long-term safety concerns. Five-year clinical trial outcomes and clinical experience have demonstrated durable virologic suppression in both treatment-naïve and treatment-experienced patients, including patients with extensive antiretroviral history and documented antiretroviral resistance. Studies have also exhibited low adverse effect rates and reliable long-term safety lending to improved tolerance. Several trials have evaluated the reduction in adverse effects in patients switched from various antiretroviral agents to RAL. Treatment-naïve studies have demonstrated a lipid-neutral effect in patients on RAL-containing regimens. When transitioning patients from a ritonavir-boosted PI regimen, statistically significant decreases in total plasma cholesterol, low-density lipoprotein, and triglycerides were demonstrated. Given its negligible interaction with the cytochrome P450 system, RAL displays minimal drug-drug interactions, making it a good option for ageing patients on multiple medications (2).

Study Design

This is an observational retrospective cohort in real world to describe RAL data, including NUC-sparing regimens, in aged HIV patients. It is a phase IV study. 90 patients will be enrolled from the Department of Public Health and Infectious Diseases of "Sapienza" University of Rome. More than 4000 HIV patients are followed at this Department of Public Health and Infectious Diseases of "Sapienza" University of Rome. More than 50% of these patients are ≥ 50 years. From 10 to 12% are treated with a raltegravir based- regimen.

In this retrospective analysis all naïve patients on raltegravir-based regimens and all patients switched to raltegravir-based regimens will be considered. For raltegravir-based regimens we mean raltegravir as third agent in a triple regimen with NRTIs and also raltegravir-based regimens in NUC-sparing therapies.

Raltegravir initiation is equivalent to baseline.

All consecutive patients fulfilling the following inclusion criteria are considered eligible:

* HIV-1 infected patients,
* aged ≥ 60 years old
* naive patients receiving raltegravir based-regimen, including Nuc-sparing regimens,
* experienced patients with virological suppression (HIV-1 RNA<50 copies) who had switched from any antiretroviral drug to raltegravir-based regimens (including Nuc-sparing regimens) because of toxicity, convenience or other reasons.

Data are collected from medical records. The Time horizon for patient follow-up for outcome is at least 12 months.

The following information will be extracted from the database of the Department:

* demographics (age, sex, race)
* smoking
* risk factors for HIV infection
* time from HIV-1 diagnosis (years)
* history of AIDS diagnosis
* hepatitis C virus (HCV) co-infection
* hepatitis B virus (HBV) co-infection
* presence of co-morbidities (including diabetes, hypertension, CVD, CKD, cancer, etc)
* reasons for switching to raltegravir
* time with HIV-1 RNA < 50 copies/mL before switch
* BMI
* Hematology (Hb, PLT)
* Creatinine
* eGFR (CKD-EPI formula)
* Phosphorus
* Calcium
* AST
* ALT
* alkaline phosphatase
* total, direct, indirect bilirubin
* proteinuria
* total, HDL-, LDL-cholesterol
* triglycerides
* glycemia
* HIV-RNA
* CD4+, CD8, CD4/CD8 ratio since the start of raltegravir
* previous ART regimen and number of previous antiretroviral agents.

Follow-up will count from the date of start of raltegravir to VF/TF or last available visit, whichever first occurred

AEs were classified as mild/moderate, severe or life threatening, according to DAIDS Classification. AEs were considered unrelated to RAL, possibly related or related, according to physician criteria.

Safety data will be descriptive; no comparison data will be analyzed.

The primary endpoint will be the description of the proportion of participants with an HIV-1 viral load < 50 copies/mL.

The secondary endpoints will be:

* Change from Baseline in CD4+ T-cell counts, CD8 cell counts, CD4/ CD8 ratio
* Proportion of subjects with laboratory alterations
* Proportion of patients with adverse events (AE), serious adverse events (SAE), also according to their severity

ELIGIBILITY:
Inclusion Criteria:

* signature of informed consent
* HIV-1 infected patients,
* aged ≥ 60 years old
* naive patients receiving raltegravir based-regimen, including Nuc-sparing regimens,
* experienced patients with virological suppression (HIV-1 RNA<50 copies) who had switched from any antiretroviral drug to raltegravir-based regimens (including Nuc-sparing regimens) because of toxicity, convenience or other reasons.

Exclusion Criteria:

- pregnancy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A sample size of 90 subjects will be enrolled, they will be produce two-sided 95% CI with the following width: when the sample proportion of patients with an HIV-1 viral load < 50 copies/mL is between 40% and 60%, the 95% CI width is 0.2, that correspond to the possible maximum width in this study. Corresponding widths are 0.17 for a sample proportion of 0.30 (or 0.70), 0.15 for a sample proportion of 0.20 (or 0.80) and 0.13 for a sample proportion of 0.10 (or 0.90) (PASS 11. NCSS, LLC. Kaysville, Utah, USA).
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2018-01-31 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
HIV-1 viral load | 12 months
  HIV-1 viral load < 50 copies/mL

SECONDARY OUTCOMES:
CD4+ T-cell counts | 12 months
  Change from Baseline in CD4+ T-cell counts (delta)
CD8 cell counts | 12 months
  Change from Baseline in CD8 cell counts (delta)
CD4/ CD8 ratio | 12 months
  Change from Baseline in CD4/ CD8 ratio (delta)

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Umberto I Hospital, Rome, Italy

REFERENCES:
- [Background] Pavone P, Giustini N, Fimiani C, Paoletti F, Falciano M, Salotti A, Di Sora F, Al Moghazi S, Mezzaroma I, Vullo V, d'Ettorre G. Long-Term Treatment With Raltegravir is Associated with Lower Triglycerides and Platelets Count in the Older HIV+ Population: Results from the Ral-Age Study. Curr HIV Res. 2017 Nov 23;15(5):355-360. doi: 10.2174/1570162X15666170927124558. PMID 28969567
- [Derived] Santinelli L, Ceccarelli G, Borrazzo C, Celani L, Pavone P, Innocenti GP, Spagnolello O, Fimiani C, Ceci F, Di Sora F, Mezzaroma I, Mastroianni CM, d'Ettorre G. Real word outcomes associated with use of raltegravir in older people living with HIV: results from the 60 months follow-up of the RAL-age cohort. Expert Rev Anti Infect Ther. 2020 May;18(5):485-492. doi: 10.1080/14787210.2020.1733415. Epub 2020 Feb 25. PMID 32096433